CLINICAL TRIAL: NCT05620550
Title: Evaluation of the Effect of Ozonated Oil on the Healing of Palatal Donor Area of Free Gingival Grafts.
Brief Title: Effect of Ozonated Oil on Healing of Palatal Area.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Elizangela Cruvinel Zuza, Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ozonated
Record Dates: First submitted 2022-10-03; First posted 2022-11-17 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Healing Surgical Wounds
Keywords: Healing; Ozone; Autografts; Oral mucosa

STUDY DESIGN:
Intervention Model Description: This is a prospective longitudinal clinical trial, being a patient-centered, double-blinded (patient and examiner), randomized by lottery, placebo-controlled study.
Who Masked: Participant, Care Provider
Masking Description: Patients will receive ramdomly one of the bottles with oil, identified as A or B. One contains sunfower ozonated oil and the other non ozonated sunflower oil. Both the patient and the operator will be blinded,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ozonated oil (Experimental): treatment of scar area with ozonated oil
  Interventions: Procedure: ozonated oil
- non ozonated oil (Sham Comparator): treatment of scar area with non ozonated oil
  Interventions: Procedure: non ozonated oil

INTERVENTIONS:
Procedure: ozonated oil — Post operative scar treatment with ozonated oil
  Arms: ozonated oil
Procedure: non ozonated oil — Post operative scar treatment with non ozonated oil
  Arms: non ozonated oil

SUMMARY:
Despite the good clinical results and advantages of using autogenous grafts, such as subepithelial connective grafts and free gingival grafts, the removal of grafts from the palate can result in greater postoperative morbidity. The objective of the present study will be to perform a clinical evaluation of the effect of ozonated oil on the healing of palatal wounds, after the removal of free gingival grafts, to be used in the post-extraction sockets, with the purpose of preserving the alveolar ridge. This is a prospective longitudinal clinical trial, being a patient-centered, double-blind, randomized by lottery, placebo- controlled study. The groups will be divided as follows: 1) EGL Group (control): after the removal of the EGL, the palatal wound will be treated with non-ozonized sunflower oil (placebo), applied once a day, for seven days. days; 2) EGL + Oz Group (test): after removal of the EGL, the palatal wound will be treated with ozonated sunflower oil with a peroxide index between 510 - 625 meq/kg (Oleozon®, São Paulo, Brazil), applied once a day, for seven days. The clinical evaluation and the healing process will be evaluated through the remaining scar area (RSA), Epithelialization (E) and Tissue Edema (TE). Assessments will be performed at baseline (after EGL removal) and at 3, 7, and 14 days. Measurement of levels of Malondialdehyde (MDA) and 4-Hydroxinonenal (4-HNE) for oxidative stress will be performed at days 3 and 7. Quality of life questionnaire (OHIP-14) and pain scale (VAS) will be applied. The data will initially be tested for normality by the Shapiro-Wilk test. If the data are parametric, Analysis of Variance (ANOVA) can be applied, but if they are non-parametric, the Kruskal-Wallis test can be applied, followed by Dunns, for comparison between groups. The significance level will be set at 5%.

DETAILED DESCRIPTION:
Study design This is a prospective longitudinal clinical trial, being a patient-centered, double-blind (patient and examiner), randomized by lottery, placebo-controlled study. The intention will be to serve patients at the dental clinics of the Nova Friburgo Health Institute, however, due to the pandemic, provisionally, until the calls return, some patients will be treated in a private dental office. Research volunteers will be attended to, complying with all biosafety procedures and will receive all care free of charge, in addition to the acrylic plate to be used after surgery, as well as all materials to be used before and after the procedure, as well as such as pain control medications.

Participants eligible for inclusion criteria will be invited to participate in the research, voluntarily, after clarifying doubts about the project and will sign an informed consent form. All principles of this study will be established in accordance with the Declaration of Helsinki. The study protocol will be analyzed and must receive approval from the research ethics committee of the health institute of Nova Friburgo-RJ, Universidade Federal Fluminense.

Sample calculation The sample calculation was performed considering the primary outcome. Considering the t test for two independent samples regarding the residual healing area in square milimetersl in the ozone group (36.04 ± 9.66) vs. control (48.21 ± 13.2) at 14 days (80% power; alpha level of 0.05), a sample of 14 patients per group was estimated. The program used to calculate the sample size was BioEstat 5.3 (Mamirauá , Belém, PA, Brazil).

Clinical groups and procedures Epithelial free gingival tissue (EGL) grafts will be removed from the palate to be placed in a post - extraction socket in order to achieve ridge preservation. Both procedures, extraction and obtaining the EGL, will be performed in the same surgical procedure. In the first surgical step, the tooth will be extracted using atraumatic instruments . In the second step, the EGL will be removed from the palate, in a standardized way, using a circular scalpel with 8 mm in diameter and 2 mm in thickness (Maximus Instrumental Odontológico®, Contagem, Brazil). The EGL will be adjusted at the entrance of the alveolus and sutured with 5.0 non-resorbable monofilament nylon thread (Ethicon ®, Johnsons & Johnsons do Brasil®, São José dos Campos, São Paulo, Brazil).

The donor area will be sutured with non-resorbable 4.0 polypropylene thread , considering that this thread is a monofilament thread , in order not to accumulate bacterial biofilm (Ethicon ®, Johnsons & Johnsons do Brasil ®, São José dos Campos, São Paulo, Brazil) . After suturing, the patient will receive a 1 mm thick acetate plate that covers part of the donor area of the palate, providing protection to the palatal wound against mechanical trauma. The suture from the palatal region will be removed at 7 days, while the suture from the recipient area will be removed at 14 days. Only the donor area will be evaluated in the present study.

The groups will be divided as follows:

* EGL group (control): after removal of the EGL, the palatal wound will be treated with non-ozonized sunflower oil (placebo), applied once a day, for seven days.
* EGL + Ozone Group (test): after EGL removal, the palatal wound will be treated with ozonized sunflower oil with a peroxide index between 510 - 625 meq /kg (Oleozon ®, São Paulo, Brazil), applied once per day for seven days.

Surgeries will be performed by a single operator, while clinical evaluations will be performed by another operator, duly trained and calibrated.

Postoperative guidelines Postoperative medication will be as follows: Amoxicillin 500 mg (1 capsule 3 times a day, for 7 days) and Dipyrone sodium 500 mg (1 tablet, every 4 hours, for 3 days only in case of pain). Dipyrone will only be recommended in case of pain and the patient should note on a specially prepared form if there was a need for consumption and the amount ingested each day.

The patient will be instructed to apply the oil provided with the aid of a cotton swab, once a day at night, after brushing the teeth, putting the acrylic plate right after to sleep. It is important to emphasize the use of the plate so that the drug has the desired effect. This card will be used for 7 days. Important not to use any mouthwash , just conventional brushing and flossing.

Clinical Evaluation Clinical evaluation and healing process will be evaluated as follows: a) remaining scar area, b) Epithelialization (E) and c) Tissue edema. Assessments will be performed at baseline (after EGL removal) and at 3, 7, and 14 days.

1. Remaining scar area (ARC): standardized photographs will be taken (brightness, distance and angle of 45º in relation to the palate), with a PCP-UNC 15 millimeter periodontal probe (Hu- Friedy ®, Chicago, Illinois, USA) being positioned to standardization in millimeters of the area to be measured in software ( Image J-NIH, Bethesda, USA). Wound area will be measured in square milimeters at, 3, 7 and 14 days after EGL removal.
2. Epithelialization (E): the wound area will be stained with an evidencing solution (Replack ® Dentisply , Pennsylvania, USA) and measured at the respective intervals, and the epithelialized area will be calculated as a percentage. Fibrin, granulation tissue and scar tissue scores: The score used was adapted from other study, considering: a) Score of the presence of a fibrin clot in: 0- presence of the entire wound extension with fibrin clot; 1- presence of ≥ 75% of fibrin clot; 2- presence of <75% to ≥ 50% of fibrin clot; 3- presence of <50% to ≥25% of fibrin clot; 4- presence of < 25% of fibrin clot; 5- absence of fibrin clot; b) Presence of granulation tissue score in: 0- absence of granulation tissue; 1- presence of < 25% of tissue; 2- presence of <50% to ≥25% of tissue; 3- presence of <75% to ≥ 50% of tissue; 4- presence of ≥ 75% of tissue; 5- presence of the entire extension with granulation tissue; c) Presence of scar tissue score in: 0- absence of scar tissue; 1- incomplete wound closure with < 25% scar tissue; 2- incomplete wound closure with <50% to ≥25% scar tissue; 3- incomplete wound closure with <75% to ≥ 50% scar tissue; 4- incomplete wound closure with ≥ 75% scar tissue; 5- complete wound closure.
3. Tissue edema (TE): the edema will be evaluated at 3 and 7 postoperative days, being considered dichotomously, as absent (0) or present.

Calibration Calibration will be performed on five patients, who will not be included in the research. The evaluator (PJ) will be trained and calibrated for ARC measurements (at baseline and 7 days after surgery) and the measurements will be performed at two different times, one week apart. The intraclass correlation will be evaluated by the BioEstat 5.0 program (Mamiraua , Pará, Brazil). Statistical significance will be set at 5%.

immunological evaluation Measurement of VEGF (vascular endothelial growth factor; pg /ml) and TGF-beta (transforming growth factor beta; pg /ml) levels in the donor region will be performed. For this, an absorbent paper tip will be used, which will be positioned in the donor area of the palate for 30 seconds, without pressure. VEGF , originally known as vascular permeability factor, is a signal protein produced by cells that stimulates blood vessel formation. TGF-beta is a protein that controls cell proliferation, differentiation and other functions in most cells. Malondialdehyde (MDA) and 4-Hydroxinonenal (4-HNE) will be evaluated for oxidative stress . The samples will be collected and placed in sterile eppendorfs , containing phosphate-buffered saline solution with 0.05% Tween 20, being stored in a freezer at -20 o C. The immunological evaluation will be performed at 3 and 7 days.

Quality of life

The instrument to assess the Oral Health-Related Quality of Life of individuals will be the questionnaire called Oral Health Impact Profile (OHIP-14). This questionnaire will only be applied on the 7th day. The seven dimensions of oral impact:

* Limitation Functional (items 1 and 2),
* Pain (items 3 and 4),
* Discomfort Psychological (items 5 and 6),
* Inability Physics (items 7 and 8),
* Inability Psychological (items 9 and 10),
* Social Disability (items 11 and 12)
* Disadvantage (items 13 and 14).

Each dimension reflects the impact of the general oral condition on certain aspects namely:

1. The Functional Limitation dimension includes questions regarding speech difficulties and reduced taste sensitivity;
2. In the Pain dimension, questions are asked about the sensation of pain experienced , as well as the discomfort in the act of eating;
3. Regarding the Psychological Discomfort dimension, the concern and stress that the oral condition may cause are explored;
4. The Physical Disability dimension refers to the possible loss of food and the need to interrupt meals;
5. In the Psychological Disability dimension, questions are asked about the difficulty in relaxing and the feeling of embarrassment related to the oral condition;
6. Regarding the Social Disability dimension, this includes questions about the impact of the oral condition on relationships with others and on the difficulty in carrying out daily activities;
7. And the Disadvantage dimension, explores the person's perception of the impact of the oral condition on their life and on the inability to carry out their activities.

The OHIP-14 consists of 14 questions, which refer to oral and general health problems that people have experienced in the last twelve months. For each question, there are five response options (never=0, hardly ever=1, occasionally=2, quite often=3, and often=4). This value is then multiplied by the weight of each question (item 1: weight = .51; item 2: weight = .49; item 3: weight = .34; item 4: weight = .66; item 5: weight = . 45; item 6: weight = .55; item 7: weight = .52; item 8: weight = .48; item 9: weight = .60; item 10: weight = .40; item 11: weight = .62; item 12: weight = .38; item 13: weight = .59; item 14: weight = .41). After adding up the scores of all the questions, the final result is obtained, which can vary between 0 and 28 points. The higher the score, the greater the impact of issues on quality of life.

Analysis of postoperative discomfort Patients were instructed to score postoperative discomfort on a 10 mm visual analogue scale (VAS), which signal the extremes of "no pain" and "extreme pain". The VAS scale must be completed by the patient, daily, until completing 7 days. The number of analgesics ingested should also be recorded during a week.

Statistical analysis The data will initially be tested for normality by the Shapiro-Wilk test. If the data are parametric, Analysis of Variance (ANOVA) can be applied, but if they are non-parametric, the Kruskal - Wallis test can be applied, followed by Dunn 's test , for comparison between groups. The significance level will be set at 5% by the BioEstat 5.0® program (Mamiraua , Pará, Brazil).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 60 years
* Good general systemic health (self-reported by the patient)
* Plaque index and gingival index <25%
* Indication of tooth extraction and preservation of the alveolar ridge
* No morphological or pathological changes in the palate

Exclusion Criteria:

* Systemic disease (e.g. diabetes with glycosylated hemoglobin >7%, cancer, HIV, chronic inflammatory diseases, etc ) and/or with any surgical contraindication
* Patients requiring antibiotic prophylaxis or who have used systemic antibiotics corticosteroids, anti- inflammatory drugs or immunosuppressants in the last three months
* Smokers,
* Patients who have had previous periodontal surgery to remove a graft in the palate area
* Pregnant or breastfeeding
* Use of medications that interfere with healing
* Patients who present oral lesions and/or in the palate region
* Total maxillary edentulism, which makes it impossible to remove the free gingival graft due to intense resorption of the alveolar ridge

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Healing | 3 months
  The primary outcome will be the remaining scar area of the palate, using a healing score, confronting clinical results with biomarkers colected from scar area.

SECONDARY OUTCOMES:
Post operative pain and discomfort | 3 months
  For secondary outcomes, the Visual Analogue Scale will be evaluated for postoperative pain and discomfort. Groups will be compared to assess if ozonated oil has a better post operative effect.

OTHER OUTCOMES:
Quality of life scores | 3 months
  Oral Health Impact Profile scores will be used to measure post operative difference between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal Fluminense, Nova Friburgo, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anzolin AP, da Silveira-Kaross NL, Bertol CD. Ozonated oil in wound healing: what has already been proven? Med Gas Res. 2020 Jan-Mar;10(1):54-59. doi: 10.4103/2045-9912.279985. PMID 32189671
- [Result] Avila-Ortiz G, Chambrone L, Vignoletti F. Effect of alveolar ridge preservation interventions following tooth extraction: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:195-223. doi: 10.1111/jcpe.13057. Erratum In: J Clin Periodontol. 2020 Jan;47(1):129. doi: 10.1111/jcpe.13212. PMID 30623987
- [Result] Dias SB, Fonseca MV, Dos Santos NC, Mathias IF, Martinho FC, Junior MS, Jardini MA, Santamaria MP. Effect of GaAIAs low-level laser therapy on the healing of human palate mucosa after connective tissue graft harvesting: randomized clinical trial. Lasers Med Sci. 2015 Aug;30(6):1695-702. doi: 10.1007/s10103-014-1685-2. Epub 2014 Nov 6. PMID 25373688
- [Result] Isler SC, Uraz A, Guler B, Ozdemir Y, Cula S, Cetiner D. Effects of Laser Photobiomodulation and Ozone Therapy on Palatal Epithelial Wound Healing and Patient Morbidity. Photomed Laser Surg. 2018 Nov;36(11):571-580. doi: 10.1089/pho.2018.4492. Epub 2018 Sep 27. PMID 30260741
- [Result] Kumar T, Arora N, Puri G, Aravinda K, Dixit A, Jatti D. Efficacy of ozonized olive oil in the management of oral lesions and conditions: A clinical trial. Contemp Clin Dent. 2016 Jan-Mar;7(1):51-4. doi: 10.4103/0976-237X.177097. PMID 27041901
- [Result] Miguel MMV, Mathias-Santamaria IF, Rossato A, Ferraz LFF, Figueiredo-Neto AM, de Marco AC, Casarin RCV, Wallet SM, Tatakis DN, Mathias MA, Santamaria MP. Microcurrent electrotherapy improves palatal wound healing: Randomized clinical trial. J Periodontol. 2021 Feb;92(2):244-253. doi: 10.1002/JPER.20-0122. Epub 2020 Aug 30. PMID 32783220
- [Result] Travagli V, Zanardi I, Valacchi G, Bocci V. Ozone and ozonated oils in skin diseases: a review. Mediators Inflamm. 2010;2010:610418. doi: 10.1155/2010/610418. Epub 2010 Jul 4. PMID 20671923
- [Result] Wessel JR, Tatakis DN. Patient outcomes following subepithelial connective tissue graft and free gingival graft procedures. J Periodontol. 2008 Mar;79(3):425-30. doi: 10.1902/jop.2008.070325. PMID 18315424